CLINICAL TRIAL: NCT07405476
Title: A Phase II Clinical Trial of Neoadjuvant Zanidatamab for HER2+ Localized Colorectal Cancer
Brief Title: Zanidatamab Before Surgery for the Treatment of HER2 Positive Colon and Rectal Cancer in Patients Planned for Curative Intent Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Olumide Gbolahan, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P012862; WINSHIP6609-25 (Other: Emory University Hospital/Winship Cancer Institute); NCI-2026-00566 (Registry Identifier: Clinical Trials Reporting Program); P30CA138292 (NIH)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colon Carcinoma; Colorectal Carcinoma; Rectal Carcinoma; Stage I Colon Cancer AJCC v8; Stage I Colorectal Cancer AJCC v8; Stage I Rectal Cancer AJCC v8; Stage II Colon Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Rectal Cancer AJCC v8; Stage III Colon Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — zanidatamab; Watchful Waiting; Observation; Radioisotopes; Cerebral Ventriculography; Endoscopy; Magnetic Resonance Spectroscopy; X-Rays; Specimen Handling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (zanidatamab, surgical resection) (Experimental): Patients receive zanidatamab IV over 90-150 minutes on day 1 of each cycle. Cycles repeat every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgical resection on study followed by adjuvant chemotherapy as per standard of care. Additionally, patients undergo echocardiography or MUGA scan, sigmoidscopy, CT or MRI, and blood sample collection throughout the study. Patients also undergo archival tissue sample collection or biopsy during screening.
  Interventions: Biological: Zanidatamab; Procedure: Resection; Other: Patient Observation; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Endoscopic Procedure; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Biopsy Procedure; Procedure: Digital Rectal Examination; Other: Electronic Health Record Review
- Cohort 2 (zanidatamab) (Experimental): Patients receive zanidatamab IV over 90-150 minutes on day 1 of each cycle. Cycles repeat every 14 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients then optionally undergo surgical resection or observation as per standard of care. Additionally, patients undergo echocardiography or MUGA scan, sigmoidscopy, CT, MRI, blood sample collection, and digital rectal exam throughout the study. Patients also undergo archival tissue sample collection or biopsy during screening.
  Interventions: Biological: Zanidatamab; Procedure: Resection; Other: Patient Observation; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Procedure: Endoscopic Procedure; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Biopsy Procedure; Procedure: Digital Rectal Examination; Other: Electronic Health Record Review

INTERVENTIONS:
Biological: Zanidatamab — Given IV
  Other Names: 2169946-15-8, Anti-HER2/HER2 Bispecific Antibody ZW25,; HER2 x HER2 Bispecific Antibody ZW25, ZANIDATAMAB, Zanidatamab-hrii, Ziihera, ZW-25, ZW25
Procedure: Resection — Undergo surgical resection
  Other Names: Resection, resection, Surgical Resection, SURGICAL RESECTION, Surgical Resection, Surgical Resection, Surgical Resection
Other: Patient Observation — Undergo observation
  Other Names: active surveillance, Active Surveillance, deferred therapy, expectant management, observation, Observation, watchful waiting, Watchful Waiting
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC, Echocardiography, Echocardiography, ECHOCARDIOGRAPHY, echocardiography, Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan, Equilibrium Radionuclide Angiography, Gated Blood Pool Imaging, Gated Heart Pool Scan, MUGA, MUGA Scan, Multi-Gated Acquisition Scan, Radionuclide; Ventriculogram Scan, Radionuclide Ventriculography, Ventriculography, RNV Scan, RNVG, SYMA Scanning, Synchronized Multigated Acquisition Scanning
Procedure: Endoscopic Procedure — Undergo sigmoidscopy
  Other Names: Endoscopic Examination, Endoscopic Procedure, Endoscopy, ENDOSCOPY, Endoscopy, Endoscopy, endoscopy, Endoscopy, ES
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT, CAT Scan, Computed Axial Tomography, Computed Tomography, Computed Tomography,; Computerized Axial Tomography, Computerized axial tomography (procedure), Computerized Tomography,; Computerized Tomography, Computerized Tomography (CT) scan, CT, CT Scan, Diagnostic CAT Scan, Diagnostic CAT Scan Service Type, tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance, Magnetic Resonance Imaging, Magnetic Resonance Imaging, Magnetic Resonance Imaging, magnetic resonance imaging,; Magnetic Resonance Imaging, Magnetic Resonance Imaging (MRI), Magnetic resonance imaging (procedure), Magnetic Resonance Imaging Scan, Medical Imaging,; Magnetic Resonance / Nuclear Magnetic Resonance, MR, MR, MR Imaging, MRI, MRI, MRI, MRI, MRI, MRI,; MRI Scan, MRI Scan, MRI Scan, MRI Scan, MRIs, NMR Imaging, NMRI, NMRI, nuclear magnetic resonance imaging, Nuclear Magnetic Resonance Imaging, sMRI, Structural MRI
Procedure: Biospecimen Collection — Undergo blood and/or archival tissue sample collection
  Other Names: Biological Sample Collection, Biological Sample Collection, Biospecimen Collected, Biospecimen Collection, Specimen Collection
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy, BIOPSY, Biopsy, Biopsy, Biopsy, biopsy, Biopsy, Biopsy, Biopsy, Biopsy, Biopsy, BIOPSY_TYPE, BIOPSY_TYPE, BIOPSY_TYPE, Bx
Procedure: Digital Rectal Examination — Undergo digital rectal examination
  Other Names: Digital Rectal Examination, digital rectal examination, DRE, DRE
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This phase II trial studies how well giving zanidatamab before surgery (neoadjuvant) works in treating patients with colon and rectal cancer that is human epidermal growth factor receptor 2 positive (HER2+ve) who are planned for curative intent treatment. Zanidatamab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the activity of neoadjuvant zanidatamab in HER2+ve (RAS wild type [RAS WT]) locally advanced colorectal cancer.

SECONDARY OBJECTIVES:

I. To determine the efficacy of neoadjuvant zanidatamab in HER2+ve (RAS WT) locally advanced colorectal cancer.

II. To determine the feasibility and safety of neoadjuvant zanidatamab in human epidermal growth factor receptor 2 positive (HER2+) locally advanced colorectal cancer.

TERTIARY/EXPLORATORY OBJECTIVE:

PRIMARY OBJECTIVE:

I. To determine the activity of neoadjuvant zanidatamab in HER2+ve (RAS wild type [RAS WT]) locally advanced colorectal cancer.

SECONDARY OBJECTIVES:

I. To determine the efficacy of neoadjuvant zanidatamab in HER2+ve (RAS WT) locally advanced colorectal cancer.

II. To determine the feasibility and safety of neoadjuvant zanidatamab in human epidermal growth factor receptor 2 positive (HER2+) locally advanced colorectal cancer.

TERTIARY/EXPLORATORY OBJECTIVE:

I. To evaluate biomarkers associated with the activity neoadjuvant zanidatamab in HER2+ (RAS WT) locally advanced colorectal cancer.

OUTLINE: HER2 positive colon cancer patients are assigned to cohort 1 and HER2 positive rectal cancer patients are assigned to cohort 2.

COHORT 1: Patients receive zanidatamab intravenously (IV) over 90-150 minutes on day 1 of each cycle. Cycles repeat every 14 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgical resection on study followed by adjuvant chemotherapy as per standard of care. Additionally, patients undergo echocardiography or multigated acquisition (MUGA) scan, sigmoidscopy, computed tomography (CT) or magnetic resonance imaging (MRI), and blood sample collection throughout the study. Patients also undergo archival tissue sample collection or biopsy during screening.

COHORT 2: Patients receive zanidatamab IV over 90-150 minutes on day 1 of each cycle. Cycles repeat every 14 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients then optionally undergo surgical resection or observation as per standard of care. Additionally, patients undergo echocardiography or MUGA scan, sigmoidscopy, CT, MRI, blood sample collection, and digital rectal exam throughout the study. Patients also undergo archival tissue sample collection or biopsy during screening.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed colon and/or rectal cancer planned for curative intent treatment at gastrointestinal clinics of Emory University's Winship Cancer Institute and collaborating centers
* Tumors must be HER2+ve (human epidermal growth factor receptor 2 [HER2] overexpression 3+ immunohistochemistry [IHC] or 2+ by IHC and positive fluorescence in situ hybridization [FISH] or HER2 amplification by next generation sequencing)
* Tumors must have RAS wildtype genotype
* Radiologically measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 50%)
* Platelet count > 100,000 cells/ ul (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Hemoglobin > 9g/dl (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Absolute neutrophil count > 1000 cells/dl (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN) (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Alanine aminotransferase (ALT) ≤ 3 × ULN (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Total bilirubin ≤ 1.5 × ULN, or ≤ 3 × ULN for participants with Gilbert's disease (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Glomerular filtration rate (GFR) > 60ml/min (based on creatine, and Cystatin C estimation where applicable) (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Adequate cardiac function with left ventricular ejection fraction of at least 50% (within 28 days of cycle 1 day 1, at the discretion of the investigator)
* Females of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* FCBP and men treated or enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 3 months after completion of study drug administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

  * A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions. This includes willingness to undergo mandatory blood sample draws for evaluation of correlatives
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

Exclusion Criteria:

* Participants with stage IV colon and rectal cancer even if curative intent resection is planned
* HER2 expression that does not meet documented inclusion criteria
* RAS mutation
* MSI-H or mismatch repair deficient rectal cancer
* Clinically significant cardiac disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension or any history of symptomatic congestive heart failure (CHF). Participants with known myocardial infarction or unstable angina within 6 months prior to expected date of cycle 1 day 1 (C1D1) are also excluded. Previous anticancer therapy-related CHF must have been ≤ grade 1 at the time of occurrence and must have completely resolved
* Participants receiving any other investigational agents or an investigational device within 28 days of administering the first dose of study drug
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in study
* Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-18 (Estimated); Study Completion 2029-12-18 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete and Major Pathologic Regression (Cohort 1) | At time of surgical resection
  For colon cancer, will evaluate the rate of complete and major pathologic regression in the surgical specimen based on the modified Dworak grading system. Will be reported as a proportion, and 95% exact binomial confidence interval. Will be estimated using the Clopper-Pearson method.
Radiologic Response (Cohort 2) | At 6 and 12 weeks
  Assessment will be by computed tomography chest, abdomen and magnetic resonance imaging of the rectum. Radiologic tumor response will be based on Response Evaluation Criteria in Solid Tumors 1.1. Will be reported as a proportion, and 95% exact binomial confidence interval. Will be estimated using the Clopper-Pearson method.
Tumor Regression Grades (Cohort 2) | At time of surgical resection
  Will be assessed in those who undergo surgical resection.

SECONDARY OUTCOMES:
Rate of Circulating Tumor Deoxyribonucleic Acid Clearance | Before cycle 1 day 1 of treatment and preoperatively for colon cancer patients or at 6 and 12 weeks for rectal cancer patients
Rate of Tumor Recurrence | At 2 years
  Will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median will be estimated using the Brookmeyer-Crowley approach.
Recurrence Free Survival | At 2 years
  Will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median will be estimated using the Brookmeyer-Crowley approach.
Incidence of Adverse Events | Up to 30 days post-discontinuation
  Safety will be determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5. Frequencies and percentages will be used to summarize safety events.
Proportion of Subjects who Complete Four Treatment Cycles (Feasibility) | Up to 3 years
  Frequencies and percentages will be used to summarize events.
Adverse Even Profile (Feasibility) | Up to 3 years
  Frequencies and percentages will be used to summarize events.
Rate of Perioperative Complications (Feasibility) | Up to 3 years
  Frequencies and percentages will be used to summarize events.

CONTACTS AND LOCATIONS:
Overall Officials: Olumide B. Gbolahan, MBBS, MSc, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States